CLINICAL TRIAL: NCT06841549
Title: Prognostic Value of FAPI Results in Acute Myocardial Infarction After Successful Coronary Primary Intervention
Brief Title: The Relationship Between FAPI Results and Myocardial Fibrosis After Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: FirstAHXiamenU-Liang
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — acute myocardial infarction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Echo-AMI: acute myocardial infarction followed by echo
- FAPI-AMI: acute myocardial infarction followed by FAPI
  Interventions: Other: FAPI

INTERVENTIONS:
Other: FAPI — FAPI is a new method to find the myocardial fibrosis under some conditions, like myocardial infarction or cardiac myopathy.
  Groups: FAPI-AMI

SUMMARY:
FAPI is a new method to discover the fibrosis of cardiac myocardium in some conditions, like myocardial infarction or cardiomyopathy. This purpose of this study is to find the relationship between FAPI results and myocardial fibrosis through some clinical serum inflammatory factors level. Meanwhile, it is the first time to provide the prognostic value of FAPI in the progression of acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria: acute myocardial infarction 1) after the successful primary intervention ;2) normal EF value; -

Exclusion Criteria: acute myocardial infarction 1) primary PCI failure; 2) EF reduced; 3) death during the hospitalization;

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute myocardial infarction after successful primary percutaneous intervention.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
MACE | the first month, the third month, the half year and the next year after acute myocardial infarction
  the target vessel failure, heart failure, repeated angina, arrhythmia and all-cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Quan W, Zhu T, Feng S, Huang X, Meng H, Du R, Zhu Z, Qu X, Li P, Cui Y, Shi K, Yan X, Zhang R, Li B. [68Ga]Ga-DOTA-FAPI-04 PET/MR in patients with acute myocardial infarction: potential role of predicting left ventricular remodeling. Eur J Nucl Med Mol Imaging. 2023 Feb;50(3):839-848. doi: 10.1007/s00259-022-06015-0. Epub 2022 Nov 3. PMID 36326870